CLINICAL TRIAL: NCT06912178
Title: Association of Sleep Quality With Pathologic Staging, Acupuncture Treatment in Patients With Chronic Atrophic Gastritis: a Cross-sectional Study
Status: Not yet recruiting | Type: Observational
Sponsor: Yi Liang (Other)
Collaborators: Zhejiang Provincial Department of Science and Technology (Unknown)
Responsible Party: Sponsor-Investigator, Yi Liang, Research Fellow, The Third Affiliated hospital of Zhejiang Chinese Medical University
Organization: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Other Study IDs: 20250303032132260
Record Dates: First submitted 2025-03-29; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Chronic Atrophic Gastritis (CAG)
Keywords: chronic atrophic gastritis; sleep quality; OLGA; OLGIM; pathologic; acupuncture; cross-sectional
MeSH Terms: conditions — Gastritis, Atrophic; Sleep Initiation and Maintenance Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum pepsinogen extracted and detected in venous blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Acupuncture — Whether or not a patient has been treated with acupuncture will be one of the exposure factors of interest in the study

SUMMARY:
In order to inform clinical treatment decisions and maximize treatment outcomes, this observational study set out to examine the relationship between pathological severity and sleep quality in patients with CAG. The idea that "if the stomach is not in harmony, you will be restless" is supported by this evidence from traditional Chinese medicine. Assessing patients' knowledge and acceptance of acupuncture therapy, determining the current general trend in CAG treatment, and assessing the initial effectiveness of acupuncture therapy in treating CAG with sleep disturbances. It is envisaged that the aforementioned investigations will aid in further refining the clinical research strategy of acupuncture and moxibustion with CAG with sleep disorders, enhance the effectiveness of treatment, and offer a more cost-effective and practical choice for treating CAG with sleep disorders.

The primary research issue is: can the traditional Chinese medical notion of "restlessness due to disharmony of the stomach" be validated in order to ascertain whether there is a correlation between pathological severity and sleep quality in patients with chronic atrophic gastritis? The pathological conditions of CAG patients were gathered based on the most recent gastroscopy report within a year, and the patients' sleep quality scores from the previous month were gathered via a questionnaire.

DETAILED DESCRIPTION:
This is a single-center, cross-sectional study

ELIGIBILITY:
Inclusion Criteria:

1. Have been diagnosed with chronic atrophic gastritis;
2. Be between the ages of 18 and 75, with no restrictions on gender;
3. Read the informed consent form, sign it, and consent to participate in this study.

Exclusion Criteria:

1. autoimmune gastritis (chronic atrophic gastritis type A);
2. patients with gastroesophageal reflux disease (GERD) as determined by endoscopy or other examinations, or patients with high-grade intraepithelial neoplasia pathologically as determined by upper gastrointestinal endoscopy and gastric mucosal biopsy;
3. patients with confirmed or unexcluded malignant tumors, particularly esophageal and gastric cancer;patients with other upper gastrointestinal pathologies, such as Barrett's esophagus or peptic ulcer;
4. additional physical, mental, psychological, or pathological conditions that may impact sleep scores, such as the use of medications for insomnia, night shifts, jet lag, major events, severe neurosis, menopausal syndrome, uncontrolled hyperthyroidism, severe diabetic peripheral neuropathy, within a month after surgical trauma, etc.
5. People who use medicines that can make you sleepy at the same time and stop using them for less than a month;
6. People who can't finish the questionnaire because they're unconscious, can't talk regularly, or have other issues; people who don't have enough information.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This multicenter clinical investigation is coordinated by Zhejiang Chinese Medical University (ZCMU) with participant enrollment conducted at the Third Affiliated Hospital of ZCMU. To establish a conclusive diagnosis for each participant, the researchers conduct an upper gastrointestinal endoscopy screening and assess serum pepsinogen levels during recruitment, subsequently identifying and continuously enrolling all eligible patients at the aforementioned hospitals until the requisite sample size is attained.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
The correlation coefficient between various pathological stages of Operative Link on Gastritis Assessment (OLGA) and Operative Link on Gastric Intestinal Metaplasia (OLGIM) and sleep quality in patients with chronic atrophic gastritis (CAG) is the main o | Gastroscopy and pathology reports within one year and sleep quality assessment within one week of participant enrollment
  General condition (age, gender, height, weight, etc.), occupation, personal and family history, Helicobacter pylori infection history, acupuncture treatment, Pittsburgh sleep quality index, serum pepsinogen index, gastroscopy results, and clinical data (OLGA and OLGIM for gastric mucosal histopathology) were among the information that the researchers gathered. The association between the histological stages of OLGA and OLGIM in stomach mucosal histopathology and the sleep quality index in CAG patients was then examined by the researchers.

SECONDARY OUTCOMES:
Acupuncture treatment response and sleep quality relationships, as well as other pertinent risk factors, were secondary outcomes | Patient's treatment to date after diagnosis of chronic atrophic gastritis, and whether participant has received acupuncture in the last 3 months
  The clinical research program of acupuncture and moxibustion with CAG with sleep disturbances was further adjusted to evaluate the relationship between acupuncture treatment and sleep quality in CAG patients. The researchers looked into how CAG patients were treated overall, including whether they had previously undergone acupuncture treatment, their preferences for different acupuncture treatments, and their willingness and acceptance of acupuncture treatment. Additionally, the quality of the CAG patients' sleep throughout the previous month was examined.

CONTACTS AND LOCATIONS:
Locations (1):
- the Ethics Board of Te Thnird Affiliated Hospital of Zhejjiang Chinese Medicinal University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF